CLINICAL TRIAL: NCT01861392
Title: Analisys of Neuromuscular Response, Postural Balance and Quality of Life of Diabetics Type 2 After Sensory-motor Training: Blind Random Controled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, PHD Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1143-3618
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus; Quality of Life; Exercise Therapy; Postural Balance
Keywords: postural balance sensory motor trayning physical therapy modalities diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Quality of Life

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sensory-motor training (Active Comparator): Guidelines + sensory-motor training.Evaluation Biomechanical data will be collected (balance, baropodometry, electromyography strength and joint position sense), as well as questionnaires ADDQoL and BESTest. The intervention will be twice a week for 45 minutes for 12 weeks, divided into three phases: heating, sensory-motor training and cool-down, with monitoring of blood pressure and blood glucose.
  Interventions: Procedure: sensorio-motor training
- guidelines (Active Comparator): receive the same guidelines and reviews that group orientation and training sensorineural engine and will be guided home exercises for postural twice a week 45 minutes for 12 weeks.
  Interventions: Procedure: sensorio-motor training

INTERVENTIONS:
Procedure: sensorio-motor training
  Other Names: quality of life

SUMMARY:
Background: The individual's ability to sustain itself in the upright position, effectively adjusting the body's movements and reacting to external stimuli, postural control strategies represent essential activities of daily living. Diabetes mellitus type 2 (DM-2) is considered a more problem of Public Health as having complications deficit in functional performance of the lower limbs and falls, which can interfere with the maintenance of balance, and is a strong predictor of functional limitations self referred. Aim: To assess quality of life and the answers neuromuscular balance and baropodometric after sensory-motor training in patients with type 2 diabetes. Method: To be recruited 50 volunteers aged between 45 to 64 years with DM-2, of both sexes, divided into two groups: 1) Guidelines and 2) Guidelines + sensory-motor training. Biomechanical data will be collected (balance, baropodometry, electromyography strength and joint position sense), as well as questionnaires ADDQoL and BESTest. The intervention will be twice a week for 45 minutes for 12 weeks, divided into three phases: heating, sensory-motor training and cool-down, with monitoring of blood pressure and blood glucose. There will be a follow up after 3 months of intervention. Statistical analysis will be used normality test to verify the data distribution and consistent statistical test for the appropriate comparisons within and between groups, and adopted a significance level of 5%. Expected Results: Considering previous studies that demonstrate improvement in postural balance static and dynamic responses under the forward training protocol sensorimotor disease Diabetes mellitus type 2, is expected to improve neuromuscular, balance, distribution plant, the joint position sense and the quality of life of voluntary DM-2.

Keywords: physical therapy modalities, exercise therapy, postural balance, Diabetes Mellitus, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus type 2 with controlled blood glucose
* Absence of skin lesions or fractures of the lower limbs in the last 6 months -Plantar malformations
* Severe postural abnormalities and limb length difference.

Exclusion Criteria:

* Use of medications that can have negative effects on the function of cognition, attention and psychomotor (ie, opioids, antiepileptics, anxiolytics, antipsychotics, hypnotics and sedatives)
* Diagnosis of cardiovascular, neurological, rheumatological and musculoskeletal disorders that may interfere with activities of daily living
* Presence of vestibular disorders

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Postural balance training diabetic type 2 | four years

SECONDARY OUTCOMES:
Quality of life of diabetics type 2 | four years

CONTACTS AND LOCATIONS:
Overall Officials: Ariane H M Pletsch, PHD Student, Principal Investigator — University of Sao Paulo; Rinaldo Roberto Jesus Guirro, PHD, Study Director — University of Sao Paulo
Locations (1):
- Rinaldo Roberto de Jesus Guirro, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Suprak DN. Shoulder joint position sense is not enhanced at end range in an unconstrained task. Hum Mov Sci. 2011 Jun;30(3):424-35. doi: 10.1016/j.humov.2011.02.003. Epub 2011 Mar 27. PMID 21444119
- [Background] Vandekerckhove M, Vermeire E, Weeren A, Van Royen P. Validation of the Diabetes Obstacles Questionnaire (DOQ) to assess obstacles in living with type 2 diabetes in a Belgian population. Prim Care Diabetes. 2009 Feb;3(1):43-7. doi: 10.1016/j.pcd.2009.02.003. Epub 2009 Mar 4. PMID 19264569
- [Background] Song CH, Petrofsky JS, Lee SW, Lee KJ, Yim JE. Effects of an exercise program on balance and trunk proprioception in older adults with diabetic neuropathies. Diabetes Technol Ther. 2011 Aug;13(8):803-11. doi: 10.1089/dia.2011.0036. Epub 2011 May 11. PMID 21561371
- [Derived] Borges NCS, Pletsch AHM, Buzato MB, Terada NAY, Cruz FMFD, Guirro RRJ. The effect of proprioceptive training on postural control in people with diabetes: A randomized clinical trial comparing delivery at home, under supervision, or no training. Clin Rehabil. 2021 Jul;35(7):988-998. doi: 10.1177/0269215521989016. Epub 2021 Jan 28. PMID 33508955
- See also: Related Info — http://www.fmrp.usp.br